CLINICAL TRIAL: NCT04260581
Title: Is Long-term Use of Amantadine Effective in Parkinson Disease?
Brief Title: Is Long-term Use of Amantadine Effective in PD?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1909-072-1064
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Amantadine; Long-term effect
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD patients who have taken amantadine (Experimental)
  Interventions: Drug: Determination of drug effects through amantadine cessation

INTERVENTIONS:
Drug: Determination of drug effects through amantadine cessation — Patients will discontinue amantadine, which has been taken since beginning of diagnosis.

SUMMARY:
The investigator aims to assess whether long-term use of amantadine is effective in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Amantadine is used in the early stages of Parkinson's disease (PD). However, amantadine is known to be relatively weak compared to other antiparkinsonian drugs such as levodopa, dopamine agonist or Mao-B inhibitor and its effects are limited in early months, so it is rarely used than other drugs.

Recently, several studies have identified the long-term effects of amantadine on dyskinesia, but the basis is still insufficient.

Therefore, this study aims to investigate the long-term effectiveness of amantadine in patients with PD. Participants who have used amantadine since the early stages of diagnosis undergo clinical evaluations including the Montreal Cognitive Assessment (MoCA), Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Freezing of Gait-Questionnaire (FOG-Q), Non-motor Symptom Scale (NMSS) and Parkinson's Disease Questionnaire-39 (PDQ-39). Then, participants stop taking amantadine. To investigate the long-term effect, clinical evaluations except MoCA are repetitively assessed at 4- and 8-week follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been taking amantadine since the beginning of diagnosis
2. Patients who have taken amantadine for more than five years
3. Patients with Parkinson's disease who are aged 40 years or older

Exclusion Criteria:

1. Patient who stops amantadine or is hypersensitive to amantadine
2. Patients who have undergone brain surgery, including deep brain stimulation
3. Patient identified as atypical parkinsonism
4. Patients with psychiatric conditions such as dementia, major depression or bipolar disorder who are difficult to assess
5. Patients who are currently unable to follow up at our hospital

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 4-week f/u in Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III score | Baseline, 4 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 132]
Change from baseline to 8-week f/u in Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III score | Baseline, 8 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 132]

SECONDARY OUTCOMES:
Change from baseline to 4-week f/u in Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I score | Baseline, 4 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 52]
Change from baseline to 8-week f/u in Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I score | Baseline, 8 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 52]
Change from baseline to 4-week f/u in Movement Disorder Society Unified Parkinson's Disease Rating Scale Part II score | Baseline, 4 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part II score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 52]
Change from baseline to 8-week f/u in Movement Disorder Society Unified Parkinson's Disease Rating Scale Part II score | Baseline, 8 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part II score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 52]
Change from baseline to 4-week f/u in Movement Disorder Society Unified Parkinson's Disease Rating Scale Part IV score | Baseline, 4 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part IV score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 24]
Change from baseline to 8-week f/u in Movement Disorder Society Unified Parkinson's Disease Rating Scale Part IV score | Baseline, 8 weeks
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part IV score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 24]
Change from baseline to 4-week f/u in Hohr and Yahr stage score | Baseline, 4 weeks
  Hohr and Yahr stage score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 5]
Change from baseline to 8-week f/u in Hohr and Yahr stage score | Baseline, 8 weeks
  Hohr and Yahr stage score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 5]
Change from baseline to 4-week f/u in Freezing of Gait Questionnaire score | Baseline, 4 weeks
  Freezing of Gait Questionnaire score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 24]
Change from baseline to 8-week f/u in Freezing of Gait Questionnaire score | Baseline, 8 weeks
  Freezing of Gait Questionnaire score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 24]
Change from baseline to 4-week f/u in Non-motor Symptom Scale score | Baseline, 4 weeks
  Non-motor Symptom Scale score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 360]
Change from baseline to 8-week f/u in Non-motor Symptom Scale score | Baseline, 8 weeks
  Non-motor Symptom Scale score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 360]
Change from baseline to 4-week f/u in Parkinson's Disease Questionnaire-39 score | Baseline, 4 weeks
  Parkinson's Disease Questionnaire-39 score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 156]
Change from baseline to 8-week f/u in Parkinson's Disease Questionnaire-39 score | Baseline, 8 weeks
  Parkinson's Disease Questionnaire-39 score will be used to determine the efficacy of amantadine. Higher scores mean a worse outcome. [minimum 0, maximum 156]

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No